CLINICAL TRIAL: NCT04887155
Title: Mobile-enhanced Transdiagnostic Group Treatment for Adolescents at Risk for Severe Mood Disorders
Brief Title: Mobile-enhanced Group CBT for Adolescents at Risk Severe Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Marc J. Weintraub, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-000036
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Adolescents; Mood Disorders
Keywords: cognitive behavioral therapy (CBT); mobile health (mHealth); Group treatment
MeSH Terms: conditions — Mood Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT)_no app (Active Comparator)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Cognitive behavioral therapy (CBT) with mobile app (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — Group-based transdiagnostic cognitive-behavioral treatment

SUMMARY:
Although cognitive-behavioral therapy (CBT) has shown efficacy in reducing symptoms and rates of mood relapse in adolescents at high risk for severe mood disorders (SMD; i.e., bipolar I/II disorder and recurrent or unremitting major depression), a significant limitation to the CBT's efficacy is the low rate of participant adherence to the prescribed between-session homework tasks. Mobile health applications have the potential to improve adherence to and acceptance of treatment through embedded treatment content, skill-practice, thought and symptom monitoring, all of which are facilitated by reward contingencies and notifications. This study examines whether a mobile application-enhanced CBT can improve participant adherence and treatment acceptance for adolescents at high risk for SMD.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-5 criteria for at least one past major depressive disorder, persistent depressive disorder, or unspecified bipolar disorder
2. Be 13-17 years old
3. English speaking and able to complete written questionnaires
4. Ability to attend pre-determined group session time(s)
5. Access to a smartphone to engage with the study app
6. Medication usage is acceptable, but not required

Exclusion Criteria:

1. Regular use or current abuse of a psychoactive drug
2. Evidence of behavioral problems that are thought to interfere with group treatment
3. Suicidality that requires more intensive treatment
4. Meeting DSM 5 criteria for bipolar I or II disorder, a psychotic disorder, or significant psychiatric symptoms (e.g., self-injurious behavior) that require more intensive treatment
5. Concurrent participation in cognitive-behavioral therapy
6. Inability to travel to study sessions and assessments

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- [Derived] Weintraub MJ, Ichinose MC, Zinberg JL, Salimian A, Brown RD, Morgan-Fleming G, Gamarra JM, Tran T, Miklowitz DJ. A randomized trial of an app-enhanced group cognitive behavioral therapy for adolescents with mood or psychotic spectrum disorders. J Consult Clin Psychol. 2025 Mar;93(3):131-143. doi: 10.1037/ccp0000946. PMID 40014504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited adolescents from two specialty outpatient programs at the UCLA Semel Institute - the Child and Adolescent Mood Disorders Program and the Center for the Assessment and Prevention of Prodromal Syndromes
Pre-assignment Details: 196 youth phone screened
  Phase I Open Trial:
  33 youth assessed 31 youth enrolled
  Phase II RCT:
  66 youth assessed 60 youth enrolled
Groups:
- Phase I Open Trial-Cognitive Behavioral Therapy (CBT) With Mobile App; Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App: The treatment delivered in this study is a modified version of the Unified Protocol (UP) for Adolescents, a CBT protocol for adolescents with emotional disorders. The treatment included nine, 90-minute weekly group sessions delivered in three modules - psychoeducation, behavioral skills, and cognitive skills.
  Participants in this conditions were also provided with access to a mobile application. The app was designed to help adolescents accomplish three treatment tasks: (1) review the treatment session content, (2) practice treatment skills, (3) and review and log their psychiatric symptoms and functional status (also known as the symptom check-in). Participants were able to review their treatment skill practice and track their symptoms in a section of the app called 'Review My Progress.' The app was used as a direct tool in the therapy session, as it was used by clinicians to review the treatment materials and have the participants practice the treatment skills in sessions. Additionally, the app served as a method to bridge sessions by allowing participants to review the prior session's content and practice treatment skills from their mobile device. The app also contained three primary engagement features: 1) text reminders to conduct weekly skill practice and symptom logging, 2) emojis that were earned upon completion of the weekly treatment skill practice, and 3) a skills streak counter indicating the consecutive weeks the participant has completed their skill practices.
- Phase II RCT-Cognitive Behavioral Therapy (CBT)_no App: The treatment delivered in this study is a modified version of the Unified Protocol (UP) for Adolescents, a CBT protocol for adolescents with emotional disorders. The treatment included nine, 90-minute weekly group sessions delivered in three modules - psychoeducation, behavioral skills, and cognitive skills.
Period: Overall Study
Arm/Group | Phase I Open Trial-Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT-Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Started | 31 | 30 | 30
Completed | 24 | 25 | 24
Not Completed | 7 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App; Phase II RCT- Cognitive Behavioral Therapy (CBT) With Mobile App: The treatment delivered in this study is a modified version of the Unified Protocol (UP) for Adolescents, a CBT protocol for adolescents with emotional disorders. The treatment included nine, 90-minute weekly group sessions delivered in three modules - psychoeducation, behavioral skills, and cognitive skills.
  Participants in this conditions were also provided with access to a mobile application. The app was designed to help adolescents accomplish three treatment tasks: (1) review the treatment session content, (2) practice treatment skills, (3) and review and log their psychiatric symptoms and functional status (also known as the symptom check-in). Participants were able to review their treatment skill practice and track their symptoms in a section of the app called 'Review My Progress.' The app was used as a direct tool in the therapy session, as it was used by clinicians to review the treatment materials and have the participants practice the treatment skills in sessions. Additionally, the app served as a method to bridge sessions by allowing participants to review the prior session's content and practice treatment skills from their mobile device. The app also contained three primary engagement features: 1) text reminders to conduct weekly skill practice and symptom logging, 2) emojis that were earned upon completion of the weekly treatment skill practice, and 3) a skills streak counter indicating the consecutive weeks the participant has completed their skill practices.
- Phase II RCT- Cognitive Behavioral Therapy (CBT)_no App: The treatment delivered in this study is a modified version of the Unified Protocol (UP) for Adolescents, a CBT protocol for adolescents with emotional disorders. The treatment included nine, 90-minute weekly group sessions delivered in three modules - psychoeducation, behavioral skills, and cognitive skills.
- Total: Total of all reporting groups
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT- Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT- Cognitive Behavioral Therapy (CBT) With Mobile App | Total
Number analyzed (Participants) | 31 | 30 | 30 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 30 | 30 | 91
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 21 | 58
  Male | 12 | 12 | 9 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 1 | 8
  White | 24 | 19 | 21 | 64
  More than one race | 2 | 3 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Depressive mood disorder diagnosis [Number; unit: Participants] — Number of Participants with a Depressive Mood Disorder Diagnosis
  Participants | 25 | 22 | 25 | 72

OUTCOME MEASURES:

1. Primary Outcome: Treatment Skill Practice
Description: Sum of all treatment skill practices completed through the course of the treatment (based on adolescent report).
Time Frame: 9-week treatment period
Measure: Mean (Standard Deviation); unit: treatment skill practices
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT-Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT- Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 24 | 24 | 25
treatment skill practices | 16.1 (8.8) | 56.2 (33.6) | 44.3 (43.6)

2. Secondary Outcome: Mobile Application Usability Scale
Description: Mobile application (app) acceptability as rated on a 5-point scale (i.e., minimum = 1, maximum = 5) with higher values indicating greater acceptability
Time Frame: Measured at the end of the 9-week treatment period
Population: No App condition did not receive the study app
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App: The treatment delivered in this study is a modified version of the Unified Protocol (UP) for Adolescents, a CBT protocol for adolescents with emotional disorders. The treatment included nine, 90-minute weekly group sessions delivered in three modules - psychoeducation, behavioral skills, and cognitive skills.
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 24 | 0 | 25
units on a scale | 3.9 (1.3) |  | 4.3 (0.8)

3. Primary Outcome: Psychosocial Treatment Compliance Scale
Description: Clinician-rated of participant overall treatment compliance. Scores range from 17-85 (17 5-point Likert scale items) with higher scores indicating greater treatment compliance.
Time Frame: 9-week treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 24 | 24 | 25
units on a scale | 64.6 (11.2) | 66.42 (10.47) | 67.83 (9.0)

4. Primary Outcome: Mobile Application Use
Description: Frequency of mobile application (app) usage within the condition that received the mobile application, ranging from 0 to unlimited maximum with higher scores indicating more app usage.
Time Frame: 9-week treatment period
Population: No App Condition did not receive the study app
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 24 | 0 | 25
units on a scale | 8.8 (7.5) |  | 9.6 (5.0)

5. Secondary Outcome: Children's Depression Rating Scale, Revised
Description: Measures depressive symptom severity. Scores range from 17-113 (14 7-point items and 3 5-point items) with higher scores indicating greater depressive severity.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The number analyzed in one or more rows differs from overall number analyzed due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 44.2 (11.7) | 45.7 (10.4) | 46.2 (11.6)
  Post-treatment: number analyzed (Participants) | 24 | 24 | 22
  Post-treatment | 36.3 (8.5) | 36.8 (11.8) | 35.9 (11.5)
  3-month follow-up: number analyzed (Participants) | 24 | 24 | 21
  3-month follow-up | 35.9 (12.0) | 33.3 (11.2) | 34.4 (14.2)

6. Secondary Outcome: Young Mania Rating Scale
Description: Measure manic symptom severity. Scores range from 0-60 (7 5-point items and 4 9-point items) with higher scores indicating greater manic severity.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 10.1 (6.1) | 10.3 (5.2) | 9.6 (5.1)
  Post-treatment: number analyzed (Participants) | 24 | 24 | 26
  Post-treatment | 9.2 (5.3) | 7.3 (5.1) | 6.0 (4.2)
  3-month follow-up: number analyzed (Participants) | 24 | 24 | 25
  3-month follow-up | 7.9 (5.2) | 6.9 (5.8) | 6.7 (4.1)

7. Secondary Outcome: Clinical Global Assessment Scale
Description: Measures overall functioning on a 1-100 scale, with higher scores indicating better functioning.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 57.9 (11.9) | 47.7 (7.4) | 44.5 (7.5)
  Post-treatment: number analyzed (Participants) | 24 | 24 | 26
  Post-treatment | 65.2 (7.0) | 54 (9.3) | 58.1 (9.8)
  3-month follow-up: number analyzed (Participants) | 24 | 24 | 25
  3-month follow-up | 67.8 (9.0) | 61.7 (14.1) | 61.7 (15.7)

8. Secondary Outcome: Clinical Global Impression
Description: Measures overall clinical functioning from 1-7, with higher scores indicating greater psychiatric severity.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 4.0 (1.2) | 4.5 (0.9) | 4.4 (0.9)
  Post-treatment: number analyzed (Participants) | 24 | 24 | 26
  Post-treatment | 3.6 (0.7) | 3.5 (1.2) | 3.4 (1.1)
  3-month follow-up: number analyzed (Participants) | 24 | 24 | 25
  3-month follow-up | 3.3 (0.9) | 3.0 (1.0) | 3.0 (1.3)

9. Secondary Outcome: Symptom Checklist 90
Description: Participant-reported psychiatry symptoms. Scores range from 0 - 360 (90 5-point Likert items) with higher scores indicating greater symptom severity.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 104.4 (76.1) | 135.0 (72.2) | 106.4 (50.8)
  End of treatment: number analyzed (Participants) | 24 | 30 | 30
  End of treatment | 100.3 (74.2) | 105.2 (85.6) | 86.5 (66.0)
  End of study: number analyzed (Participants) | 24 | 24 | 25
  End of study | 71.0 (77.2) | 87.6 (72.6) | 84.2 (64.6)

10. Secondary Outcome: Difficulties With Emotion Regulation
Description: Participant reported their difficulties with emotion regulation. Scores range from 36 - 180 (36 5-point items) with higher scores indicating greater distress.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 106.0 (23.0) | 101.9 (28.6) | 99.5 (18.7)
  End of treatment: number analyzed (Participants) | 24 | 30 | 30
  End of treatment | 103.22 (26.8) | 97.7 (31.5) | 90.9 (21.7)
  End of study: number analyzed (Participants) | 24 | 24 | 25
  End of study | 87.0 (26.1) | 92.2 (28.7) | 89.9 (17.4)

11. Secondary Outcome: KINDL
Description: Quality of life measure. Scores range from 0 - 120 (30 5-point items) with higher scores indicating better quality of life.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population total between rows is due to study participant attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
units on a scale
  Baseline | 105.7 (10.9) | 90.63 (15.2) | 95.13 (9.97)
  End of treatment: number analyzed (Participants) | 24 | 30 | 30
  End of treatment | 104.4 (9.8) | 97.3 (13.1) | 97.5 (16.7)
  End of study: number analyzed (Participants) | 24 | 24 | 25
  End of study | 109.5 (10.7) | 102.3 (15.1) | 100 (18.2)

12. Secondary Outcome: Depression Anxiety & Stress Scale
Description: Parent reported mood, anxiety and stress. Scores range from 0 - 63 (21 4-point items) with higher scores indicating greater distress.
Time Frame: Measured prior to treatment (0 months), at the end of the 9-week treatment, and the end of the 21-week study period.
Population: The difference between the analysis population totals between rows is due to participant attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
Number analyzed (Participants) | 31 | 30 | 30
score on a scale
  Baseline | 20.5 (14.9) | 12.97 (8.0) | 11.7 (11.3)
  End of treatment: number analyzed (Participants) | 24 | 30 | 30
  End of treatment | 19.2 (16.2) | 12.5 (7.2) | 11.5 (7.1)
  End of study: number analyzed (Participants) | 24 | 24 | 25
  End of study | 15.0 (15.8) | 11.8 (9.7) | 11.0 (9.3)

ADVERSE EVENTS:
Time Frame: 21-weeks (i.e., from enrollment through completion of 21-week study)
Arm/Group | Phase I Open Trial - Cognitive Behavioral Therapy (CBT) With Mobile App | Phase II RCT - Cognitive Behavioral Therapy (CBT)_no App | Phase II RCT - Cognitive Behavioral Therapy (CBT) With Mobile App
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Most of the adolescents were diagnosed with a depressive spectrum disorder. Ratings of skill practice were made based on adolescent and clinician report, but there was no definitive method of confirming skill practice completion in the standard UP group, nor was there any examination of the proficiency/quality of skill practice across both conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04887155/Prot_SAP_000.pdf